CLINICAL TRIAL: NCT00248235
Title: Randomized Controlled Trial of Progressive Resistance Exercise Training for Spinal Accessory Neurapraxia/ Neurectomy in Head and Neck Cancer Survivors
Brief Title: Resistance Exercise Training for the Shoulder and Neck Following Surgery for Head and Neck Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HN-4-0023
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Neoplasms
Keywords: exercise; rehabilitation; head and neck neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- PRET (Experimental): Progressive Resistance Exercise Training: upper extremity 6-8 exercises
  Interventions: Behavioral: Exercise
- Standard Care (Active Comparator): Standard Care: physical therapy - range of motion, 6-8 strengthening exercises
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
The purpose of this study is to investigate the effect of a progressive therapeutic exercise program on specific physical and functional deficits in the neck and shoulder region occurring as a result of head and neck cancer treatment.

DETAILED DESCRIPTION:
We will be conducting a randomized controlled trial to evaluate the effects of progressive resistance exercise training (PRET) on shoulder and neck dysfunction due to spinal accessory neurapraxia/ neurectomy in patients with head and neck cancer. Sixty-four head and neck cancer survivors will be randomly assigned to PRET or standard care. Participants assigned to the PRET group will exercise 3 times per week for 12 weeks. The goal of the exercise program will be to enhance scapular stability, and improve mobility and strength of the upper extremity. The resistance exercise program will be progressive in terms of the number of sets and repetitions performed, as well as amount lifted, depending on baseline strength levels and overall performance status. The primary outcomes for the study include pain and dysfunction, active and passive range of motion measures, strength and endurance testing, and quality of life. Nerve conduction testing and electromyography will be performed to assess/ monitor the status of the spinal accessory nerve and trapezius muscle function respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx OR squamous cell carcinoma metastatic to the neck from unknown primary site; probable occult mucosal origin in the head and neck
2. Surgical treatment includes radical neck dissection, modified radical neck dissection and other variants of functional/selective neck dissection
3. Karnofsky Performance Status greater than or equal to 60%
4. No evidence of residual cancer in the neck and no distant (M0) metastasis
5. Participants must have completed their head and neck cancer treatment

Exclusion Criteria:

1. A history of shoulder or neck pathology unrelated to cancer treatment
2. Serious co-morbid medical illness or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pain and dysfunction (baseline, 12 weeks, 6 months, 12 months) | baseline, 12 weeks, 6 months, 12 months
Active and passive range of motion (baseline, 12 weeks) | baseline, 12 weeks
Muscular strength and endurance (baseline, 12 weeks) | baseline, 12 weeks
Quality of life (baseline, 12 weeks, 6 months, 12 months) | baseline, 12 weeks, 6 months, 12 months

SECONDARY OUTCOMES:
Anxiety, depression and fatigue (baseline, 12 weeks, 6 months, 12 months) | baseline, 12 weeks, 6 months, 12 months
Nerve conduction testing (baseline, 12 weeks as indicated) | Baseline
Electromyography (baseline, 12 weeks as indicated) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — Professor, Faculty of Physical Education and Recreation, University of Alberta
Locations (1):
- Behavioral Medicine Laboratory, University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] McNeely ML, Parliament M, Courneya KS, Seikaly H, Jha N, Scrimger R, Hanson J. A pilot study of a randomized controlled trial to evaluate the effects of progressive resistance exercise training on shoulder dysfunction caused by spinal accessory neurapraxia/neurectomy in head and neck cancer survivors. Head Neck. 2004 Jun;26(6):518-30. doi: 10.1002/hed.20010. PMID 15162353